CLINICAL TRIAL: NCT03238118
Title: Randomized Clinical Trial Comparing Attention Bias Modification, Attention Control and Psychoeducation for Irritability in Children and Adolescents
Brief Title: Attention Bias Modification, Attention Control and Psychoeducation for Irritability in Children and Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 39602514700005327
Record Dates: First submitted 2017-08-01; First posted 2017-08-03 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Irritability
Keywords: irritability; severe mood dysregulation; disruptive mood dysregulation disorder

STUDY DESIGN:
Intervention Model Description: A) The first sub-group (n=60) will participate in the intervention group (the attention bias modification training) and will receive psychoeducation; B) The second sub-group (n=60 children) will participate in the attention control condition and will receive psychoeducation; C) The third sub-group (n= 20) will receive only psychoeducation. Children will be randomly assigned to one of these three groups. Both children and parents will be blind to group assignment.
  Parents will provide written informed consent for children's participation. This study was approved by the Ethics Committee of Hospital de Clinicas de Porto Alegre.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants and caregivers will be blinded to the intervention and control groups. They will not be blinded to the psychoeducation group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Attention bias modification training (Experimental): For attention-toward-positive, stimuli are colour-pictures of 16 angry and 16 happy faces (half female). Each happy face is presented 10 times, and each angry face presented 80 times across trials, balanced across the different positions in the 3 × 3 matrix. This yielded 160 training trials (two blocks of 80 trials). Children had to mouse-click on the happy face within the 3 × 3 matrix of angry faces as quickly and as accurately as possible. The matrix disappeared after the child mouse-clicked on the correct face and the next trial began.
  Interventions: Other: Attention bias modification training; Other: Psychoeducation
- Attention Control Training (Placebo Comparator): For attention-training-control, stimuli are 20 colour-pictures of individual birds and flowers used in prior visual-search tasks with children. Children mouse-clicked on the bird presented amongst flowers as quickly and accurately as possible. Other task parameters were similar to the attention-toward-positive task (160 training trials). No performance feedback is given in either condition.
  Interventions: Other: Attention Control Training; Other: Psychoeducation
- Psychoeducation (Placebo Comparator): Psychoeducation is an intervention that is characterized by informing the participant of their irritability symptoms. The goal is to teach participants how to understand their symptoms, explain their treatment modalities, recognize signs that may lead to a possible crisis, and provide tips and strategies on how to deal with irritability.
  Interventions: Other: Psychoeducation

INTERVENTIONS:
Other: Attention bias modification training — Participants will complete the assigned attention-training task three times a week for two weeks (six sessions), yielding 960 trials. Each session consists of three parts: evaluating the individual baseline, training and testing. Participants will also be required to complete a self-report assessment before and after each session. Participants will be evaluated at baseline, the end of week 1 and at the end of week 2 by blind investigators.
  Psychoeducation Participants will receive psychoeducation once a week for two weeks. Participants will also be required to complete a self-report assessment before and after each session of psychoeducation. Participants will be evaluated at baseline, the end of week 1 and at the end of week 2 by blind investigators.
  Arms: Attention bias modification training
Other: Attention Control Training — Attention Control Training Participants will complete the assigned attention-training task three times a week for two weeks (six sessions), yielding 960 trials. Each session consists of three parts: evaluating the individual baseline, training and testing. Participants will also be required to complete a self-report assessment before and after each session. Participants will be evaluated at baseline, the end of week 1 and at the end of week 2 by blind investigators.
  Psychoeducation Participants will receive psychoeducation once a week for two weeks. Participants will also be required to complete a self-report assessment before and after each session of psychoeducation. Participants will be evaluated at baseline, the end of week 1 and at the end of week 2 by blind investigators.
  Arms: Attention Control Training
Other: Psychoeducation — Participants will receive psychoeducation once a week for two weeks. Participants will also be required to complete a self-report assessment before and after each session of psychoeducation. Participants will be evaluated at baseline, the end of week 1 and at the end of week 2.

SUMMARY:
The aim of this project is to evaluate the efficacy of an attention bias modification training if compared to an attention control and psychoeducation to reduce the symptoms of irritability among children with high levels of irritability.

DETAILED DESCRIPTION:
Children with high levels of irritability have showed significant bias towards threatening faces. Computerized training programs have showed to be able to successfully modify these biases in children with mood and anxiety disorders. Of particular importance, a study examined the effects of attention training towards positive stimuli on attention biases and anxiety symptoms in pediatric anxiety disorders. In the attention-towards-positive condition, children searched picture arrays for a happy face amongst angry faces. In the attention-training control condition, children searched for a bird amongst flowers. This study showed significantly greater reductions in clinician-rated diagnostic severity and number of diagnoses of anxiety with that training. However, no study has investigated the role of these training in children and adolescents with high levels of irritability The present project, aims to examine the effects of the attention bias modification training and compare to attention-training control condition and psychoeducation in children with high levels of irritability.

ELIGIBILITY:
Inclusion Criteria:

* children aged 9 to 12 years with symptoms of irritability who scored above the 90% percentile for their existing symptoms on Affective Reactivity Index

Exclusion Criteria:

* a diagnosis of intellectual disability.

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2020-09-24 (Actual); Study Completion 2020-09-24 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline to endpoint in the "Irritability Subscale" of The Multidimensional Assessment of Preschool Disruptive Behavior (mean values) | two weeks
  The Multidimensional Assessment of Preschool Disruptive Behavior is a developmentally sensitive questionnaire, which is used to assess temper loss in terms of tantrum features and anger regulation. A total of 39 items are rated in terms of frequency over the past month: 0 = Never in the past month; 1 = Rarely (less than weekly); 2 = Some days (1-3 days per week); 3 = Most days (4-6 days); 4 = Daily; and 5 = Multiple times per day.

SECONDARY OUTCOMES:
Mean change from baseline to endpoint in the Affective Reactivity Index | two weeks
  The Affective Reactivity individual items are scored 0,1, 2, and only the first six items are summed to form the total score - the seventh is an impairment item and it is analyzed separately.
Mean change from baseline to endpoint in The Extended Strengths and Weaknesses Assessment of Normal Behavior | two weeks
  The Extended Strengths and Weaknesses Assessment of Normal Behavior has been developed in order to capture variance associated with both strengths and weaknesses to generate a near-normal distribution in epidemiological samples. For each of the 30 items, evaluators assess how well the child handles emotions and behaves compared to other children of the same age - far below average, below average, slightly below average, about average, slightly above average, above average and far above average.

OTHER OUTCOMES:
Anxiety: The parent- and child-report formats of the Spence Children's Anxiety Scale | two weeks
  The Extended Strengths and Weaknesses Assessment of Normal Behavior has been developed in order to capture variance associated with both strengths and weaknesses to generate a near-normal distribution in epidemiological samples. For each of the 30 items, evaluators assess how well the child handles emotions and behaves compared to other children of the same age - far below average, below average, slightly below average, about average, slightly above average, above average and far above average.
Depression: Mood and Feelings Questionnaire | two weeks
  The Mood and Feelings Questionnaire is a 33-item questionnaire based on "Diagnostic and Statistical Manual of Mental Disorders" (DSM)-III-R criteria for depression. Consists of a series of descriptive phrases regarding how the subject has been feeling or acting recently. Codings reflect whether the phrase was descriptive of the subject most of the time, sometimes, or not at all in the past two weeks.
Attention-Deficit/Hyperactivity Disorder: The Multimodal Treatment Study for Attention-Deficit/Hyperactivity Disorder Swanson - Version IV | two weeks
  The items from the DSM-IV (1994) criteria for Attention-Deficit/Hyperactivity Disorder are included for the two subsets of symptoms: inattention (items 1-9) and hyperactivity/impulsivity (items 11-19). Also, items are included from the DSM-IV criteria for Oppositional Defiant Disorder (items 21-28) since it often is present in children with Attention-Deficit/Hyperactivity Disorder.
Profile of Mood State | two weeks
  The Profile of Mood State contains 65 adjectives rated by participants on a 5-point scale. Six factors are derived that include tension, depression, anger, fatigue, vigor and confusion.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Salum, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Paola Paganella Laporte, Porto Alegre, Rio Grande do Sul, Brazil